CLINICAL TRIAL: NCT04946266
Title: Prospective Validation of the Prognostic Value of Long Non-coding MFI2-AS1 RNA in Localized Clear Cell Kidney Cancers
Acronym: MFI2-PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7349
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical intervention — Surgical intervention with collection of tissue material

SUMMARY:
An exploratory analysis of the expression of MFI2-AS1 will be performed at the plasma level with the objective of comparing this expression with tumor tissue. The objective would be to be able to use long non-coding RNA as a biomarker for diagnosis before tissue analysis and for patient follow-up. In addition, correlations will be made between tumor expression of MFI2-AS1 and genetic and immune alterations in tumors in order to better clarify the link between the expression of this long non-coding RNA and the characteristics of the tumor and of the tumor. tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Localized kidney tumors> T1a
* Patient having signed an informed consent
* Patient affiliated to a health insurance plan
* Subject having signed a consent form to participate in research and the constitution of a collection and genetic analyzes

Exclusion Criteria:

* Metastatic carcinoma from the outset
* Contraindication to performing a TAP CT with injection of contrast product
* Inability to provide informed information about the subject (subject in an emergency situation, difficulties in understanding, etc.)
* Subject under legal protection
* Subject under tutorship or curatorship
* Pregnancy
* Feeding with milk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with localized kidney tumors
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Expression of MFI2-AS1 | 36 month
  To assess the link between tumor expression of MFI2-AS1 in patients with localized clear cell kidney carcinoma and the occurrence of relapse

CONTACTS AND LOCATIONS:
Overall Officials: TRICARD Thibault, Principal Investigator — les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided